CLINICAL TRIAL: NCT05532709
Title: Comparative Effects of Plyometric and Circuit Training on Speed, Agility and Power in Volleyball Players
Brief Title: Effects of Plyometric and Circuit Training in Volleyball Players
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/22/0404
Record Dates: First submitted 2022-09-05; First posted 2022-09-08 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Volleyball Players
MeSH Terms: interventions — Plyometric Exercise; Circuit-Based Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plyometric training (Experimental): The plyometric training program progressed from level one (weeks one and two; 1-2 sets of 10 repetitions) to level two (weeks three and four; 1-2 sets of 8 repetitions) and finally level three (weeks five and six; 1-2 sets of 6 repetitions). Plyometric training programs included both leg jumps, single-leg jumps, hurdle jumps, drop jumps, box jumps or lunge jumps
  Interventions: Other: Plyometric training
- circuit training (Experimental): The circuit training consists of 6 exercises, divided in 2 blocks (1st block contains
  ½ squats, bench press and pushups and 2nd block contains burpees, squat thrust and lunges) of 3 minutes.
  Interventions: Other: Circuit training

INTERVENTIONS:
Other: Plyometric training — m level one (weeks one and two; 1-2 sets of 10 repetitions) to level two (weeks three and four; 1-2 sets of 8 repetitions) and finally level three (weeks five and six; 1-2 sets of 6 repetitions). Plyometric training programs included both leg jumps, single-leg jumps, hurdle jumps, drop jumps, box jumps or lunge jumps
  Arms: Plyometric training
Other: Circuit training — The circuit training consists of 6 exercises, divided in 2 blocks (1st block contains
  ½ squats, bench press and pushups and 2nd block contains burpees, squat thrust and lunges) of 3 minutes.
  Arms: circuit training

SUMMARY:
Circuit training is a formed type of training in which the trainees goes through a series of selected exercises of activities that are performed in a sequence or in a circuit. Plyometric training is an intense, advanced form of exercise in which the muscles are first stretched, then contracted (the pre-stretching makes the muscle contract with greater force). Plyometric training is one of the most popular training approaches adopted by coaches and strength and conditioning professionals in both, team and individual sports.

DETAILED DESCRIPTION:
Circuit training is a formed type of training in which the trainees goes through a series of selected exercises of activities that are performed in a sequence or in a circuit. Plyometric training is an intense, advanced form of exercise in which the muscles are first stretched, then contracted (the pre-stretching makes the muscle contract with greater force). Plyometric training is one of the most popular training approaches adopted by coaches and strength and conditioning professionals in both, team and individual sports. This study will be a randomized clinical trial and will be conducted in Pakistan sports complex. Non-probability convenience sampling technique will be used to collect the data. The sample size of total 28 athletes will be taken in this study. The participants will be divided into two groups: group I will follow plyometric training and group II will receive circuit training. The plyometric training program progressed from level one (weeks one and two; 1-2 sets of 10 repetitions) to level two (weeks three and four; 1-2 sets of 8 repetitions) and finally level three (weeks five and six; 1-2 sets of 6 repetitions). Plyometric training programs included both leg jumps, single-leg jumps, hurdle jumps, drop jumps, box jumps or lunge jumps.

The circuit training consists of 6 exercises, divided in 2 blocks (1st block contains

½ squats, bench press and pushups and 2nd block contains burpees, squat thrust and lunges) of 3 minutes. Cooper's test, Sprint test, Vertical jump test and Agility shuttle run test will be used to evaluate the results after 6 weeks

ELIGIBILITY:
Inclusion Criteria:

* Only Males
* Age between 16-25 years
* volleyball players
* Players have spent at least one year in sports EXCLUSION CRITERIA
* Players undergone surgery or had an accident.
* Any malignant or chronic diseases
* Patients with infections or any inflammatory disease
* Patients with contraindications to exercise therapy (uncontrolled hypertension, respiratory diseases.
* Patients with spinal deformities or fractures.

Ages: 16 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Cooper's test | 8 week
  The Cooper 12 minute run is a popular maximal running test of aerobic fitness, in which participants try and cover as much distance as they can in 12 minutes. purpose: to test aerobic fitness (the ability of the body to use oxygen to power it while running)
Sprint test | 8 week
  Sprints are used to primarily test an athlete's acceleration. Max speed is directly linked to initial acceleration so testing sprint times at smaller initial intervals give a picture of whether training is improving acceleration and therefore max speed.
Vertical jump test | 8 week
  The Vertical Jump test is designed to measure an applicant's lower body strength. The applicant then crouches and using the arms and legs jumps as high as possible extending the dominant arm.
  Upon reaching the top of the jump the applicant must tap the gauge "fins" to mark the jump height.
AGILITY SHUTTLE RUN TEST | 8 Week
  The 30 foot (9.15m) Agility Shuttle Run is a test of agility, in which the participant runs back and forth between two parallel lines as fast as possible, picming up blocks of wood, for a total of 120 ft. There is a similar metric version of this test, the 4x10m agility run.

CONTACTS AND LOCATIONS:
Overall Officials: Amna Shahid, t-DPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan sports board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No